CLINICAL TRIAL: NCT03981965
Title: Impact of FOCUS Guidelines on Adherence to Physical Activity in Ageing Women.
Brief Title: FOCUS Guidelines and Adherence to Physical Activity in Ageing Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Antonio Cano Sanchez, Full Professor Obstetrics and Gynecology, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FOCUS_Valencia
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Frail Elderly Syndrome; Mood; Quality of Life; Cognitive Decline; Social Interaction; Adherence, Patient
Keywords: physical activity; adherence; Frailty; Mood; Socialisation; Quality of life; Cognition
MeSH Terms: conditions — Cognitive Dysfunction; Patient Compliance; Motor Activity; Frailty | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Three groups were designed for a 24 week duration of the study. Two groups performed physical activity in two 12-week periods. A health professional acted as a supervisor during the first period. The second period was autonomous, with women providing mutual support through whatsapp, a mobile phone based social network. The first group followed the guidelines emanated from the FOCUS European project. The third group was an inactive control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focus guidelines (Experimental): Participants enrolled in a 2-phase physical activity program divided in 2 phases as described above. Briefly, The activity consisted in a 1-h set of exercises twice per week. The first 12-week phase was performed in group under the direct supervision of a health monitor. The second 12-week phase was autonomous, and consisted of the same physical performance while maintaining virtual link through a social network based on the mobile phone.
  The FOCUS guidelines provided 2 features, the participation in monthly health talks provided by the principal investigator and the availability of a virtual mailbox to transmit any comment or suggestion.
  Interventions: Other: Physical activity
- Active group (Active Comparator): Participants enrolled in a 2-phase physical activity program divided into 2 phases as described above. This group lacked the monthly talks and did not have access to the virtual mailbox.
  Interventions: Other: Physical activity
- Inactive (No Intervention): Women of similar clinical characteristic who did not participate in the PA program.

INTERVENTIONS:
Other: Physical activity — Physical activity as described previously.
  Arms: Active group; Focus guidelines

SUMMARY:
The study aimed at assessing whether the guidelines from the European project FOCUS had an effect on adherence to a physical activity program in older women. The program consisted of two 12-week periods, in which women followed a set of pre-specified exercises (1 hour, twice per week). The first period was supervised by a monitor while the second was autonomous. Support groups, in which the contact between participants was established through information and communication technologies (social-network through the mobile phone), were set up to maintain engagement between participants. Women were randomized to three arms consisting of 2 intervention groups, with and without the FOCUS guidelines, and a sedentary control. Secondary outcomes included a battery of dimensions affecting physical performance, psychological status, and quality of life.

DETAILED DESCRIPTION:
The objectives of the study consisted of assessing i) whether the use of the Guidelines derived from the European project FOCUS had an effect on the adherence to a physical activity (PA) program (primary objective), and ii) the effect of the program, which included 2 h/week of PA, on a group of dimensions related with general health, frailty, psycho-cognitive parameters, and quality of life (QoL) (secondary objectives).

The study comprised 24 weeks in which a group of 90 postmenopausal women were randomised to three arms, two in which participants were performing PA, and one control (no intervention).

The first PA group followed the FOCUS guidelines, in which women received monthly health talks and had an internet mailbox to facilitate contact with health professionals.

The PA program consisted of a twice per week 1-hour session along 24 weeks. This period was divided into two parts, a first supervised phase in which women followed group sessions under direct supervision of a monitor, and a second period in which the groups of women followed the same exercise pattern, but autonomously. A mobile phone support system (social network whatsapp) was used for inter-connection and mutual support during the autonomous period. Assessments were performed at baseline and then at 12 weeks and 24 weeks, representing the completion of the supervised and the autonomous periods, respectively.

ELIGIBILITY:
Inclusion Criteria:

Community living postmenopausal women capable of performing the physical activity program and with ability to sign the informed consent.

Exclusion Criteria:

Physical or psychological deficiencies incapacitating subjects to participate in the established physical program.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Adherence: Level of adherence to the program as assessed by attendance to the physical activity sessions. | 6 months
  Attendance will be measured as a percentage of the total number of sessions.

SECONDARY OUTCOMES:
Frailty: changes in frailty as assessed by the Fried index | 6 months
  Changes in frailty as assessed by the Fried index, which has 5 dimensions and describes a robust state (negative for all the three criteria) in addition to the pre-frail (positive for 1 or 2 criteria) and frail (positive at least in 3 criteria) status.
Cognitive function | 6 months
  Measures as per ACE-III questionnaire
Mood status | 6 months
  Measures as per HAD questionnaire
Social activities | 6 months
  Measures as per Saint Louis questionnaire
Psychological well-being as measured by the 52-item Ryff scale | 6 months
  The Ryff scale includes 52 items designed to measure six constructs of psychological well-being: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Higher total scores indicate higher psychological well-being. Respondents rate statements on a scale of 1 to 6, where 1 indicates strong disagreement and 6 indicates strong agreement.
Sleep quality, measured as per Athens Insomnia scale | 6 months
  The Athens scale aims at assessing the insomnia symptoms in individuals with sleep disorders. The scale measures 8 factors, which are intended to measure nocturnal sleep (5 factors) and daytime sleep-related disorders. Factors are rated from 0 till 3 and the cumulative score gives the final outcome. A cut-off score of 6 or higher is considered equivalent to the diagnosis of insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cano Sánchez, MD, Principal Investigator — University of Valencia
Locations (1):
- Hosp Clinico Universitario-INCLIVA, Valencia, Spain